CLINICAL TRIAL: NCT05857787
Title: Validation of Educational Effect of Nerve Tracking Function Mounted on the Ultrasound: A Randomized Comparative Trial
Brief Title: Validation of Educational Effect of Nerve Tracking Function Mounted on the Ultrasound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University (Other)
Responsible Party: Principal Investigator, Jeeyoun Moon, Professor, Seoul National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-161-1416
Record Dates: First submitted 2023-04-23; First posted 2023-05-15 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Healthy
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With nerve track function(group A) (Active Comparator): trained in the live demo method with nerve track function
  Interventions: Device: Ultrasound with nerve track function
- Without nerve track function(group B) (Active Comparator): trained in the existing live demo method without nerve track function
  Interventions: Device: Ultrasound without nerve track function

INTERVENTIONS:
Device: Ultrasound with nerve track function — The nerve track function installed in some ultrasound devices is software that accumulates ultrasound data obtained from humans and uses ultrasound to identify the target nerve through deep learning. Well-trained pain physicians use this feature to educate subjects before seeking brachial plexus and median nerve.
  Arms: With nerve track function(group A)
Device: Ultrasound without nerve track function — The nerve track function installed in some ultrasound devices is software that accumulates ultrasound data obtained from humans and uses ultrasound to identify the target nerve through deep learning. Well-trained pain physicians use ultrasound alone without this feature to educate subjects before seeking brachial plexus and median nerve.
  Arms: Without nerve track function(group B)

SUMMARY:
The purpose of this study is to find out whether the nerve track function is helpful in distinguishing appropriate anatomical structures for beginners using ultrasound.

DETAILED DESCRIPTION:
2nd, 3rd, 4th year medical school students and 1st, 2nd, 3rd year residents of anesthesiology who voluntarily signed a consent form for participation in the study are investigated for the history of previous ultrasound use and other details of the subjects before the lecture and ultrasound practice.

Well-trained pain physicians provides anatomical education on the brachial plexus supraclavicular level and the median nerve at wrist level. At this time, an ultrasound cross-sectional image of the corresponding nerve is provided. After anatomical education, research subjects (students and residents) are randomly assigned to group A or B after receiving basic education in a 1:1 ratio.

Subjects receive training for about 10 minutes to find the brachial plexus (supraclavicular level) and median nerve (carpal tunnel level) through a live demo method that directly uses ultrasound. At this time, group A receives training in the live demo method with the nerve track function, and group B receives training in the live demo method without the nerve track function.

After a 5-minute intermission, both groups A and B were asked to find the brachial plexux and median nerve without the nerve track function in the instructor's left upper limb. Each nerve is to be found within 5 minutes, and it is considered a failure after 5 minutes.

After activating the nerve track function in both groups without intermission, the educator shows the nerves corresponding to the brachial plexus at supracalvicualr level and median nerve at wrist level in the left upper limb, and conducts the same 5-minute training on finding them.

After a 5-minute intermission, with the nerve track function turned off again, ask the educator to find the brachial plexus and median nerve in the right arm.

ELIGIBILITY:
Inclusion Criteria:

* 2nd, 3rd, 4th year students at Seoul National University College of Medicine
* 1st, 2nd, 3rd year residents of anesthesiology at Seoul National University Hospital
* Those who voluntarily consented

Exclusion Criteria:

* Those who have previously identified the brachial plexus at supraclavicular level and median nerve at wrist level using ultrasound

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2024-04-23 (Estimated); Study Completion 2024-06-10 (Estimated)

PRIMARY OUTCOMES:
Success rate (%) of accurately locating a nerve in the first round in groups A and B | 5 minutes after starting to find the nerve using ultrasound
  The subjects search for the median nerve and brachial plexus after ultrasound live demo training according to the group. If each nerve is found within 5 minutes, it is considered a success.

SECONDARY OUTCOMES:
Success rate (%) of accurately locating a nerve in the second round in groups A and B | 5 minutes after starting to find the nerve using ultrasound
  After completing a first round of finding nerves, the subjects are trained using the nerve track function common to both groups, and are then asked to find nerves again. It is considered a success if each nerve is found within 5 minutes.
Subjects' assessment of the educational effect of the nerve track function | 5 minutes after the second round of finding nerves
  After completing all the procedures, the subjects expressed their satisfaction with the educational effect of nerve track function on a 5-point Likert scale. Participants will be asked to use a 5-point Likert scale, ranging from 1 to 5, for their responses. Regarding the assessment of nerve track function, the scale is explained as follows: 1 point representing "not at all helpful", 2 point representing "slightly helpful", 3 point representing "neutral", 4 point representing "somewhat helpful", and 5 point representing "very helpful".
Medical students and anesthesiology residents success rate (%) | 5 minutes after starting to find the nerve using ultrasound at first round and second round
  Among the subjects, the success rate was calculated by dividing the students of the medical school and the residents of the department of anesthesiology. Similarly, finding a nerve within 5 minutes is considered a success. Each round is calculated separately.

CONTACTS AND LOCATIONS:
Overall Officials: Jee Youn Moon, MD, PhD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhatia A, Brull R. Review article: is ultrasound guidance advantageous for interventional pain management? A systematic review of chronic pain outcomes. Anesth Analg. 2013 Jul;117(1):236-51. doi: 10.1213/ANE.0b013e31828f5ee4. Epub 2013 Apr 16. PMID 23592606
- [Background] Narouze SN, Provenzano D, Peng P, Eichenberger U, Lee SC, Nicholls B, Moriggl B; American Society of Regional Anesthesia and Pain Medicine; European Society of Regional Anaesthesia and Pain Therapy; Asian Australasian Federation of Pain Societies. The American Society of Regional Anesthesia and Pain Medicine, the European Society of Regional Anaesthesia and Pain Therapy, and the Asian Australasian Federation of Pain Societies Joint Committee recommendations for education and training in ultrasound-guided interventional pain procedures. Reg Anesth Pain Med. 2012 Nov-Dec;37(6):657-64. doi: 10.1097/AAP.0b013e318269c189. PMID 23080347
- [Background] Bodenham AR. Editorial II: Ultrasound imaging by anaesthetists: training and accreditation issues. Br J Anaesth. 2006 Apr;96(4):414-7. doi: 10.1093/bja/ael032. No abstract available. PMID 16549625
- [Background] Mendiratta-Lala M, Williams T, de Quadros N, Bonnett J, Mendiratta V. The use of a simulation center to improve resident proficiency in performing ultrasound-guided procedures. Acad Radiol. 2010 Apr;17(4):535-40. doi: 10.1016/j.acra.2009.11.010. Epub 2010 Jan 25. PMID 20097583
- [Background] Kwon SY, Hong SH, Kim ES, Park HJ, You Y, Kim YH. The Efficacy of Lumbosacral Spine Phantom to Improve Resident Proficiency in Performing Ultrasound-Guided Spinal Procedure. Pain Med. 2015 Dec;16(12):2284-91. doi: 10.1111/pme.12870. Epub 2015 Aug 3. PMID 26234900
- [Background] van Eerd M, Patijn J, Sieben JM, Sommer M, Van Zundert J, van Kleef M, Lataster A. Ultrasonography of the cervical spine: an in vitro anatomical validation model. Anesthesiology. 2014 Jan;120(1):86-96. doi: 10.1097/ALN.0000000000000006. PMID 24141229
- [Background] McVicar J, Niazi AU, Murgatroyd H, Chin KJ, Chan VW. Novice performance of ultrasound-guided needling skills: effect of a needle guidance system. Reg Anesth Pain Med. 2015 Mar-Apr;40(2):150-3. doi: 10.1097/AAP.0000000000000209. PMID 25642909